CLINICAL TRIAL: NCT03619473
Title: Standard Motorcycle Child Safety Helmet Initiative Program for the Safety of Child Pillion Riders in Malaysia
Brief Title: Standard Motorcycle Child Safety Helmet Initiative (MCHI) Program
Acronym: MCHI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universiti Putra Malaysia (Other)
Collaborators: Halliburton Foundation USA (Other); Safe Kids Worldwide USA (Unknown)
Responsible Party: Principal Investigator, Assoc Prof Dr Kulanthayan K.C. Mani, Executive Director, Universiti Putra Malaysia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: Motorcycle Child Helmet Study; 6384400 (Other Grant/Funding Number: Halliburton Foundation USA)
Record Dates: First submitted 2018-07-12; First posted 2018-08-08 (Actual); Last update posted 2018-08-08 (Actual); Status verified 2018-08

CONDITIONS: Head Injuries
Keywords: standard motorcycle child safety helmet; chinstrap; toy/game helmet
MeSH Terms: conditions — Craniocerebral Trauma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention (Experimental): the group
  1. assessed for proper helmet usage (type, chinstrap, standard helmet usage)
  2. evaluated for the behavioral of helmet usage
  3. underwent the educational session under helmet initiative program
  4. received one standard motorcycle child safety helmet per family
  5. assessed for proper helmet usage (type, chinstrap, standard helmet usage) 3 months after educational session and after received standard motorcycle child safety helmet
  6. evaluated for the behavioral of helmet usage 3 months after educational session and after received standard motorcycle child safety helmet
  Interventions: Behavioral: Standard motorcycle child safety helmet
- control (No Intervention): the group
  1. assessed for proper helmet usage (type, chinstrap, standard helmet usage)
  2. evaluated for the behavioral of helmet usage
  3. assessed for proper helmet usage after 3 months 4 evaluated for the behavioral of helmet usage after 3 months
  do not receive any educational session or standard motorcycle child safety helmet

INTERVENTIONS:
Behavioral: Standard motorcycle child safety helmet — Educational session followed by demonstration on
  * proper helmet wearing
  * how to differentiate non-standard and standard helmets
  * how to keep motorcycle safe using ABCD concept
  * importance of wearing bright clothes
  * police summon for not wearing helmets
  * live demo on poor performance of non-standard helmet
  * giving away standard motorcycle child safety helmets
  * oath taking by parents and children
  * distribution and placement of VEM on parents' motorcycles
  Arms: intervention

SUMMARY:
The main aim of this intervention study is to test the hypothesis if helmet initiative program will significantly increase helmet usage in primary school students. The secondary aim of this intervention is to evaluate the behavioral change in standard child safety helmet usage among the parent/adult riders. The study was conducted in 23 primary school in Selangor from 1st January 2016 to 31st December 2018 in three different phases.

DETAILED DESCRIPTION:
In Malaysia, the road traffic plans estimated that the number of death on road traffics might increase almost 23% from 2014-2020 (Royal Police of Malaysia, 2017). The main road crash involved the motorcyclist and the main cause of death was due to the severe head injuries. Previous study in Malaysia had reported only 20% of proper helmet usage among the adult riders (Malaysian Institute of Road Safety Research, 2015). This highlights the need to transfer the knowledge to the parent/adult riders on the importance, proper usage and availability of the standard child safety helmet and hence increase the prevalence of standard helmet usage for the pillion riders especially for the children.

ELIGIBILITY:
Inclusion Criteria:

* primary school students from selected school
* aged 7 - 12 years old
* Travel to school by motorcycle.
* the adult rider able to speak/read Malay and English

Exclusion Criteria:

* Students who are travelling to school using mode of transport other than motorcycle.
* pre school students

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2000 (Estimated)
Dates: Start 2016-01-01 (Actual); Primary Completion 2018-11-30 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
There will be increase in the prevalence of standard motorcycle child safety helmet usage in post intervention compared to pre-intervention | through study completion, an average of 1 year
  1. There will be increase in the prevalence of standard motorcycle child safety helmet usage among primary school students after the educational session under helmet initiative program as well as after the distribution of standard motorcycle child safety helmets.
  2. The educational session under helmet initiative program will provide important information about the risks of riding without standard helmet include the severity of injury to children. This will be an effective effort for continuous usage of standard helmet among child pillion riders
  3. Distribution of standard motorcycle child safety helmets will be able to increase the ownership of standard child helmet especially among those who; hence will increase the prevalence of standard motorcycle child safety helmet usage

SECONDARY OUTCOMES:
There will be increase in the prevalence of proper standard motorcycle safety helmet usage in post intervention compared to pre-intervention | through study completion, an average of 1 year
  Wearing a properly fitted, safety-approved motorcycle helmet will able to reduce head injuries.
  The educational session under helmet initiative program will provide important information about the severity of injury to children due to improper helmet usage. This will be an effective effort to reduce the prevalence of head injuries among child pillion riders
There will be increase in mean score of parents' knowledge measured using questionnaire in standard motorcycle child safety helmet usage in post intervention compared to pre-intervention | through study completion, an average of 1 year
  1. The usage of standard child motorcycle helmet among child pillion riders will be more successful when they receive consistent messages from their parents.
  2. The educational session under helmet initiative program will provide important information on the law, proper usage, risk of non-usage and the consequences to the parents which further will develope a positive attitude toward helmet wearing for children.
  3. parents' practice in helmet usage will significantly motivates the children to wear a helmet

CONTACTS AND LOCATIONS:
Locations (2):
- Malaysia (2):
  - Primary Schools in Hulu Langat District, Hulu Langat, Selangor
  - Primary Schools in Petaling Perdana District, Shah Alam, Selangor

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kulanthayan S, Umar RS, Hariza HA, Nasir MT, Harwant S. Compliance of proper safety helmet usage in motorcyclists. Med J Malaysia. 2000 Mar;55(1):40-4. PMID 11072489
- See also: safekids malaysia facebook page — https://www.facebook.com/safekidsmalaysia/